CLINICAL TRIAL: NCT01820364
Title: Phase II, Multi-center, Open-label Study of Single-agent LGX818 Followed by a Rational Combination With Agents After Progression on LGX818, in Adult Patients With Locally Advanced or Metastatic BRAF V600 Melanoma
Brief Title: LGX818 in Combination With Agents (MEK162; BKM120; LEE011; BGJ398; INC280) in Advanced BRAF Melanoma
Acronym: LOGIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn due to scientific and business considerations.
Sponsor: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLGX818X2102; 2012-004798-17 (EudraCT Number)
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Melanoma
Keywords: open-label study; BRAF inhibitor; LGX818; MEK1620; MAPK1/2 inhibitor; Pi3K inhibitor; FGFR; c-Met; CDK4/6; metastatic melanoma; BRAF; V600
MeSH Terms: conditions — Melanoma | interventions — encorafenib

ARMS (1):
- LGX818 single agent (Experimental): Patients had to have written documentation of a BRAFV600 mutation, which was to have been obtained locally on a fresh tumor biopsy (preferred) or on the most recent archival tumor sample available.
  Interventions: Drug: LGX818

INTERVENTIONS:
Drug: LGX818 — BRAF inhibitor. LGX818 was administered QD orally on a daily schedule (21-day cycles) as a flat-fixed dose and not by body weight or body surface area. LGX818 100 mg capsules and 50 mg capsules.
  Other Names: encorafenib

SUMMARY:
The primary purpose of the Phase II CLGX818X2102 study is to assess the anti-tumor activity of LGX818 in combination with selected agents.

DETAILED DESCRIPTION:
This is a phase II two part multi-center, open-label study. Part I: LGX818 single agent treatment until progression Part II: Combination treatments of LGX818 + MEK162, or BKM120, or BGJ398, or INC280, or LEE01 to assess the clinical efficacy, to further evaluate the safety of the drug combinations in patients with locally advanced or metastatic BRAF mutant melanoma after relapse on LGX818, and to determine the maximum tolerated dose of the combinations (when not established previously). These drug combinations are selected and assigned to patients based on documentation of molecular resistance mechanism.

Patients with BRAF mutant melanoma treated by LGX818 single agent in other studies can be enrolled directly in Part II of CLGX818X2102 after relapse.

Dose-escalations in the combination arms for which no MTD has been established will be based on the recommendations of a Bayesian logistic regression model guided by an escalation with overdose control criterion.

After careful evaluation of slow enrollment and the BRAF-mutant melanoma treatment landscape, recruitment was permanently halted on 26-Jul-2014.

This recruitment halt was not a consequence of any safety concern and patients who were ongoing in the study continued to be treated as per protocol.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced or metastatic melanoma
* confirmed BRAF V600 mutation
* patients naïve to a selective BRAF inhibitor
* fresh tumor biopsy at baseline, and patient agrees for a mandatory biopsy at the time of relapse
* life expectancy ≥ 3 months
* World Health Organization (WHO) Performance Status ≤ 2.

Exclusion Criteria:

* Previous treatment with RAF-inhibitor
* Symptomatic or untreated leptomeningeal disease
* Symptomatic brain metastases.
* Known acute or chronic pancreatitis
* Clinically significant cardiac disease
* AST/SGOT and ALT/SGPT > 2.5 x ULN, or > 5 x ULN if liver metastases are present
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral interventional drug
* Previous or concurrent malignancy.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation

Specific exclusion criteria for each treatment arm:

LGX818/MEK162:

History or current evidence of retinal disease History of Gilbert's syndrome.

LGX818/BKM120:

Patients with diabetes mellitus requiring insulin treatment Patient has mood disorders

LGX818/BGJ398:

History and/or current evidence of ectopic mineralization/ calcification Current evidence of corneal disorder/ keratopathy Patients with current evidence of endocrine alteration of calcium/phosphate homeostasis.

History of congenital long QT- syndrome and/or hypokalaemia CTCAE Grade ≥ 3 and/or magnesium levels below the clinically relevant lower limits before study entry.

Ionized (i) calcium (Ca) > ULN Serum inorganic phosphorus (Pi) > ULN

LGX818/LEE011 History of congenital long QT- syndrome and/or hypokalaemia CTCAE Grade ≥ 3 and/or magnesium levels below the clinically relevant lower limits before study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Array BioPharma, Study Director — 303-381-6604
Locations (6):
- Sarah Cannon Research Institute Onc Dept, Nashville, Tennessee, United States
- Novartis Investigative Site, East Melbourne, Victoria, Australia
- Novartis Investigative Site, Edmonton, Alberta, Canada
- Novartis Investigative Site, Heidelberg, Germany
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began on 04-Nov-2013 (First Subject First Visit) to the CLGX818X2102 (LOGIC 1) study. A total of 15 subjects were enrolled. The last subject's last visit occurred on 23-Mar-2015.
  Not completed subjects represents subjects that stopped treatment early, due to the corresponding reason.
Pre-assignment Details: After careful evaluation of slow enrollment and the BRAF-mutant melanoma treatment landscape, recruitment was permanently halted on 26-Jul-2014.
  This recruitment halt was not a consequence of any safety concern and patients who were ongoing in the study continued to be treated as per protocol.
Groups:
- Part I: LGX818 - Single Agent: Subjects in Part I of the study received LGX818 as a single agent.
- Part II: CLGX818 + MEK162: As per the original study design, Part II was to have five arms corresponding to the five potential combination treatments; however, only one patient was treated in this part of the study and received LGX818 in combination with MEK162.
Period: Part I: LGX818
Arm/Group | Part I: LGX818 - Single Agent | Part II: CLGX818 + MEK162
Started | 15 | 0
Completed | 1 | 0
Not Completed | 14 | 0
Not completed — Death | 1 | 0
Not completed — Administrative Problems | 3 | 0
Not completed — Adverse Event | 6 | 0
Not completed — Disease Progression | 4 | 0
Period: Part II: LGX818 + MEK162
Arm/Group | Part I: LGX818 - Single Agent | Part II: CLGX818 + MEK162
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Study Termination | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population for Baseline Demographics is composed of the Full Analysis Set, which consists of all patients who received at least one dose of LGX818.
Arm/Group | Part I: LGX818 - Single Agent
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (16.53)
Gender [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 2
  Australia | 3
  Switzerland | 6
  Germany | 1
  Spain | 3
Weight [Mean (Standard Deviation); unit: kilograms] | 80.3 (19.11)
Height [Mean (Standard Deviation); unit: centimeters] | 171.8 (9.51)
WHO/ ECOG performance status [Number; unit: participants] — Categories:
  * 0 - Fully active, able to carry on all pre-disease performance without restriction
  * 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  * 2 - Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours
  * 3 - Capable of only limited self-care, confined to bed or chair more than 50% of waking hours
  * 4 - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  participants
    0 | 14
    1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response (Overall Response Rate) Per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 (Part I & Part II)
Description: Response Evaluation Criteria In Solid Tumors (RECIST) is a set of published rules that define the status of tumors in cancer patients during a specific treatment.
  The Overall Response Rate was calculated according to the RECIST criteria, as per investigator assessment.
  Per RECIST guidelines:
  * Complete Response (CR) is the Disappearance of all target lesions.
  * Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions.
  * Progressive Disease (PD) is the at least a 20% increase in the sum of diameters of target lesions.
  * Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Baseline through study completion (approximately 2 years)
Population: This analysis is comprised of the Full Analysis Set, which consists of all patients who received at least one dose of LGX818.
Measure: Number; unit: participants
Arm/Group | Part I: LGX818 - Single Agent | Part II: CLGX818 + MEK162
Number analyzed (Participants) | 15 | 1
participants
  Complete Response | 1 | 0
  Partial Response | 8 | 0
  Progressive Disease | 1 | 1
  Stable Disease | 2 | 0
  Unknown | 3 | 0

2. Secondary Outcome: Incidence of Dose Limiting Toxicities (DLTs) (Part II)
Description: Incidence of DLTs in Part II of the study was not evaluated due to an inadequate number of patients enrolled in Part II prior to the permanent recruitment halt of this study.
Time Frame: Baseline through study completion (approximately 2 years)
Arm/Group | Part II: CLGX818 + MEK162
Number analyzed (Participants) | 0

3. Secondary Outcome: Plasma Concentration and Derived Pharmacokinetic Parameters
Description: Assessment of pharmacokinetic (PK) parameters and plasma concentration was not done due to an inadequate number of patients enrolled in Part II prior to the permanent recruitment halt of this study.
Time Frame: Baseline through study completion (approximately 2 years)
Arm/Group | Part I: LGX818 - Single Agent | Part II: CLGX818 + MEK162
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Tumor Response (Overall Response Rate) Via Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 (Part I)
Description: as for outcome 1
Time Frame: Baseline through completion of Part I of the study (approximately 2 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Part I: LGX818 - Single Agent
Number analyzed (Participants) | 15
participants
  Complete Response | 1
  Partial Response | 8
  Progressive Disease | 1
  Stable Disease | 2
  Unknown | 3

5. Secondary Outcome: Tumor Response (Overall Response Rate) Via Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 (Part II)
Description: Response Evaluation Criteria In Solid Tumors (RECIST) is a set of published rules that define the status of tumors in cancer patients during a specific treatment.
  The Overall Response Rate was calculated according to the RECIST criteria, as per investigator assessment.
  Per RECIST guidelines:
  * Complete Response (CR) is the Disappearance of all target lesions.
  * Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions.
  * Progressive Disease (PD) is the at least a 20% increase in the sum of diameters of target lesions.
  * Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  One patient with documented PD at study Day 146 entered into Part II of the study and received combination treatment of LGX818 450 mg plus MEK162 45 mg for two weeks. The patient experienced disease progression on Day 22 of Part II and discontinued the study.
Time Frame: Entry to Part II of the study through study completion (approximately 22 days)
Population: This analysis group is comprised of the Full Analysis Set, which consists of all patients who received at least one dose of LGX818.
Measure: Number; unit: participants
Arm/Group | Part II: CLGX818 + MEK162
Number analyzed (Participants) | 1
participants
  Complete Response | 0
  Partial Response | 0
  Progressive Disease | 1
  Stable Disease | 0
  Unknown | 0

6. Secondary Outcome: Molecular Status of Markers Relevant to the RAP/MEK/ERK and PI3K/AKT Pathways
Description: Molecular status was not evaluated due to an inadequate number of patients enrolled in Part II prior to the permanent recruitment halt of this study.
Time Frame: Baseline and at progression with LGX818 single agent treatment
Arm/Group | Part I: LGX818 - Single Agent | Part II: CLGX818 + MEK162
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs), Serious Adverse Events (SAEs), and Non-serious AEs were collected throughout the duration of the study, approximately 2 years. An AE was defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occur after patient's signed informed consent has been obtained. This analysis group is the Safety Set, which is all patients from the Full Analysis Set who had at least one post-baseline safety assessment.
Description: Due to slow enrollment, the study was terminated on 26-July-2014, at which time 15 patients were enrolled of Phase I of the study. The last patient last visit date occurred on 23-March-2015.
  One patient with documented PD at study Day 146 entered into Part II of the study and received combination treatment of LGX818 450 mg plus MEK162 45 mg for two weeks. The patient experienced disease progression on Day 22 of Part II and discontinued the study.
Arm/Group | Part I: LGX818 - Single Agent
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: LGX818 - Single Agent (N=15)
Hypotension (Vascular disorders) | 1
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Panic Attack (Psychiatric disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: LGX818 - Single Agent (N=15)
Flushing (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Blepharal Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyogenic Granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fatigue (General disorders) | 9
Asthenia (General disorders) | 4
Oedema Peripheral (General disorders) | 3
Face Oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 1
Menstruation Irregular (Reproductive system and breast disorders) | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1
Dyspnoea (Reproductive system and breast disorders) | 2
Procedural Pain (Injury, poisoning and procedural complications) | 1
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1
Gamma-Glutamyltransferase Increased (Investigations) | 2
Alanine Aminotransferase Increased (Investigations) | 1
Amylase Increased (Investigations) | 1
Blood Alkaline Phosphatase Increased (Investigations) | 1
Blood Cholesterol Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 1
Electrocardiogram Qt Prolonged (Investigations) | 1
Haemoglobin Increased (Investigations) | 1
Lipase Increased (Investigations) | 1
Weight Decreased (Investigations) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Long Qt Syndrome (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 5
Leukocytosis (Blood and lymphatic system disorders) | 2
Eosinophilia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Headache (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 3
Aphasia (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Hypogeusia (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
VIIth Nerve Paralysis (Nervous system disorders) | 1
Insomnia (Nervous system disorders) | 10
Cataract (Eye disorders) | 1
Conjunctival Hyperaemia (Eye disorders) | 1
Ophthalmoplegia (Eye disorders) | 1
Vision Blurred (Eye disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gingival Bleeding (Gastrointestinal disorders) | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Inguinal Hernia (Gastrointestinal disorders) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Tongue Coated (Gastrointestinal disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 10
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 9
Dry Skin (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 3
Rash Papular (Skin and subcutaneous tissue disorders) | 2
Granuloma Skin (Skin and subcutaneous tissue disorders) | 1
Palmar Erythema (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 1
Skin Hypertrophy (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Decreased Appetite (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Anal Abscess (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1
Oral Candidiasis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
Recruitment halted on 26-Jul-2014, which led to small numbers of subjects analyzed. This recruitment halt was not a consequence of any safety concern and patients who were ongoing in the study continued to be treated as per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of the sponsor's agreements with its investigators may vary. However, the sponsor does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in the clinical trial.